CLINICAL TRIAL: NCT03449316
Title: Inhaler Technique Education in Elderly Patients With Asthma or COPD: Impact on Disease Exacerbations - a Protocol for a Single-blinded Randomised Controlled Trial
Brief Title: Inhaler Technique in Elderly Patients: Impact on Disease Exacerbations
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aveiro-Aradas Family Health Unit (Other)
Responsible Party: Principal Investigator, Tiago Maricoto, Principal Investigator, Aveiro-Aradas Family Health Unit
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol V3
Record Dates: First submitted 2018-02-13; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Asthma; COPD
Keywords: Nebulizers and Vaporizers
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Two arms single blinded randomised controlled trial with a 1 year follow up
Who Masked: Outcomes Assessor
Masking Description: Blinding for the investigator that acess outcomes, that will not be involved in the intervention process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaler technique education (Experimental): This group will receive a structured and regular follow-up plan, with education on inhaler technique. Patients will be trained by a Family Doctor (the primary investigator) in terms of the inhaler technique using placebo devices similar to their own devices. A teach-to-goal approach will be used, repeating all correct steps as many times as needed in order for patients to perform them correctly at each evaluation. There will be visits at baseline and after 3, 6 and 12 months to assess outcomes. In each visit, and prior to the main intervention with the primary investigator, assessment of the inhaler technique and application of all questionnaires (clinical control, treatment adhesion and quality of life) will be performed by a secondary blinded investigator.
  Interventions: Behavioral: Inhaler technique education
- Usual Care (No Intervention): This group will receive usual care from their own Family doctors, with no specific intervention. Each doctor will perform the necessary consultations according to his real life judgment. Besides this, this group will perform visits at baseline and after 3, 6 and 12 months to assess secondary outcomes. At each visit, assessment of the inhaler technique and application of all questionnaires (clinical control, treatment adhesion and quality of life) will be performed by a secondary blinded investigator. At any appointment, if the patient asks for or if the clinician decides to teach inhaler technique, that will be recorded.
  If any adjustments are made in drug classes or device types in every participants, this information will be recorded.

INTERVENTIONS:
Behavioral: Inhaler technique education — Teaching of inhalers use with placebo devices in real training
  Arms: Inhaler technique education

SUMMARY:
Introduction COPD and Asthma affect more than 10% of the population. Most patients use their inhaler incorrectly, mainly the elderly, thereby becoming more susceptible to poor clinical control and exacerbations. Placebo device training is regarded as one of the best teaching methods, but there is scarce evidence to support it as the most effective one to improve major clinical outcomes. Our objective is to perform a single-blinded RCT to assess the impact of this education tool in these patients.

Methods and Analysis A multicentre single-blinded RCT will be set, comparing a placebo-device training programme versus usual care, with a one-year follow-up, in elderly patients with Asthma or COPD. Intervention will be provided at baseline, and after 3 and 6 months, with interim analysis at an intermediate time point. Exacerbation rates were set as primary outcomes, and quality of life, adherence rates, clinical control and respiratory function were chosen as secondary outcomes. A sample size of 146 participants (73 in each arm) was estimated as adequate to detect a 50% reduction in event rates. Two-sample proportions Chi-squared test will be used to study primary outcome and subgroup analysis will be carried out according to major baseline characteristics.

Discussion The investigators expect to confirm that inhaler performance education will significantly reduce exacerbation rate and improve clinical and functional control.

Ethics and dissemination:

Every participant will sign a consent form. A Data Safety Monitoring Board will be set up to evaluate data throughout the study and to monitor stop earlier criteria. Identity of all participants will be protected. Results will be presented in scientific meeting and published in peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of COPD or Asthma, medicated with any kind of inhaler device (pressurized Metered Dose Inhaler (pMDI) with or without Spacer, Dry Powder Inhaler (DPI) or Soft Mist), aged ≥65 years and being a regular user of primary health care services (defined as having at least one consultation performed in the last two years with his/her own Family Doctor). In order to minimize diagnostic inaccuracy, Asthma and COPD diagnosis will be reviewed in every participant at baseline prior to enrolment and according to GINA and GOLD strategies.

Exclusion Criteria:

* Severe or acute illness (such as unstable cardiovascular status, unstable angina, recent myocardial infarction (within one month) or pulmonary embolism, haemoptysis of unknown origin, recent pneumothorax (within one month), recent thoracic, abdominal or eye surgery (within one month), acute nausea or vomiting, severe respiratory distress, dementia). Patients with intermittent asthma, as well as COPD patients with mild obstruction (GOLD class I) will be excluded, since these patients do not need to take inhaler medication on a daily basis, and tend to have a low frequency of disease exacerbations.

Ages: 65 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Elderly patients
Enrollment: 146 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Evaluation at 12 months.
  This outcome will be quantifyed as "time to event"
  For Asthma, an event will be defined as increased respiratory clinical symptoms leading the patient to search for medical care, and resulting in any of the following:
  * Need for increased inhaled corticosteroid dose of at least 4x the regular dose
  * Need for increase of short-acting β2 agonists on a daily basis
  * Need for oral corticosteroids
  * Need for oral antibiotics
  * Hospitalization or Emergency Room (ER) visit with increased respiratory clinical symptoms.
  For COPD, an event will be defined as increased respiratory clinical symptoms inducing the patient to search for medical care, and resulting in any of the following:
  * Need for increase of long-acting β2 agonists on a daily basis
  * Need for oral corticosteroids
  * Need for oral antibiotics
  * Hospitalization or ER visit with increased respiratory clinical symptoms. Respiratory-related mortality and all-cause mortality will also be considered an adverse event.

SECONDARY OUTCOMES:
Clinical assessment | Evaluation at 12 months
  COPD Assessment Tools (CAT) [scale from 0 (worst) to 40 (best) points]
Clinical assessment | Evaluation at 12 months
  modified Medical Research Council (mMRC) [scale from 0 (best) to 4 (worst) points]
Clinical assessment | Evaluation at 12 months
  Control of Allergic Rhinitis and Asthma Test (CARAT) [scale from 0 (worst) to 30 (best) points]
Clinical assessment | Evaluation at 12 months
  Asthma Control Test (ACT) [scale from 5 (worst) to 25 (best) points]
Quality of Life | Evaluation at 12 months.
  Asthma Quality of Life Questionnaire (AQLQ) [scale from 32 (worst) to 224 (best) points]
Quality of Life | Evaluation at 12 months.
  St. George's Respiratory Questionnaire [scale from 0 (best) to 75 (worst) points]
Quality of Life | Evaluation at 12 months.
  Clinical COPD Questionnaire (CCQ) [scale from 0 (best) to 60 (worst) points]
Functional control | Evaluation at 12 months.
  Functional control using FEV1 in liters.
Functional control | Evaluation at 12 months.
  Functional control using FVC in liters.
Functional control | Evaluation at 12 months.
  Functional control using PEF in liters/sec.
Functional control | Evaluation at 12 months.
  Functional control using MEF25-75, in % of predicted values.
Functional control | Evaluation at 12 months.
  Functional control using FEV1/FVC ratio.
Adherence rate | Evaluation at 12 months.
  Adherence rate using the Brief Medication Questionnaire [scale from 0 (best) to 11 (worst) points]
Inhaler technique performance | Evaluation at 12 months.
  Number of errors in inhaler technique (that will be standardized to a score up to 100% scale) [To evaluate inhaler technique performance with each device, the Aerosol Drug Management Improvement Team (ADMIT) protocols and guidelines will be used, evaluating all the recommended steps for inhaler use on each one of them. For those devices that do not have any protocol from the ADMIT group, investigators will use the recommendations from the manufacture's Summary of Product Characteristics.

IPD SHARING:
Plan to Share IPD: Undecided
All data from the trial will be kept in a safe place of the principal investigator's institutional facilities and by the Data Safety Monitoring Board, in accordance with the national and international clinical research policies.

REFERENCES:
- [Derived] Maricoto T, Correia-de-Sousa J, Taborda-Barata L. Inhaler technique education in elderly patients with asthma or COPD: impact on disease exacerbations-a protocol for a single-blinded randomised controlled trial. BMJ Open. 2019 Jan 28;9(1):e022685. doi: 10.1136/bmjopen-2018-022685. PMID 30696670